CLINICAL TRIAL: NCT03154632
Title: Effectiveness of Digital Capacitive Diathermy Versus Ultrasound on Myofascial Trigger Points
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad San Jorge (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 01/2017
Record Dates: First submitted 2017-05-02; First posted 2017-05-16 (Actual); Last update posted 2018-05-03 (Actual); Status verified 2017-05

CONDITIONS: Muscle Tonus
Keywords: Myofascial trigger point; Trapezius Muscle; Diathermy; Ultrasound
MeSH Terms: conditions — Fever | interventions — Ultrasonic Therapy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- US Group (Active Comparator): Ultrasound Therapy
  Interventions: Device: Ultrasound Therapy
- DCD Group (Active Comparator): Digital Capacitive Diathermy Therapy
  Interventions: Device: Digital Capacitive Diathermy Therapy

INTERVENTIONS:
Device: Ultrasound Therapy — Ultrasound equipment will be used, choosing a continuous mode, with a frequency of 1MHz and an intensity of 1.0 W/cm2. The technique will be applied during 6 minutes with circular movements and a speed of approximately between 2.5 and 4 centimeters per second.
  Arms: US Group
Device: Digital Capacitive Diathermy Therapy — The DCD equipment will be used choosing the "musculotendinous injury FAST" program which lasts 6 minutes. The applicator will move with a velocity approximately between 2.5 and 4 centimeters per second.
  Arms: DCD Group

SUMMARY:
The main objective:

To compare the effect on muscle tone between the application of digital capacitive diathermy and the application of ultrasound on the myofascial trigger points (MTP) of the upper trapezius muscle.

Hypothesis:

The application of digital capacitive diathermy on myofascial trigger points of the trapezius muscle compared to the application of ultrasound produces objective changes in muscle tone, and this change is superior to the changes generated by the US.

DETAILED DESCRIPTION:
It is a simple-blinded randomized crossover clinical trial where volunteer subjects, older than 18 years, have a latent or active proximal MTP1 (intermediate part of the anterior margin of the upper part of the muscle near the vertical fibers of the muscle attached to clavicle) in the upper trapezius.

It will assess if there are changes in the muscle tone of the trapezius muscle after applying digital capacitive diathermy (DCD) or ultrasound (US) in the latent or active MTP1 of the trapezius muscle in healthy adults.

Each patient will receive a single session of each treatment in the affected trapezius. The order in which treatments are received - US followed by digital capacitive diathermy, or vice versa - is determined at random.

To remove any carryover of effects, there will be a week of washing period between the two interventions.

Intervention:

- DCD: The patient is positioned in prone position on stretcher. Firstly, it will apply almonds oil on the MTP1 of the upper trapezius affected. Then, it will put the "musculotendinous injury FAST" program which lasts 6 minutes; and, it will move the ultrasound applicator in contact with the skin with a velocity approximately between 2.5 and 4 centimeters per second.

- US: The patient is positioned in prone position on the stretcher. Firstly, it will select parameters (frequency: 1MHz, intensity: 1.0 W/cm2, mode: continuous). Then it will apply a slow technique of circular movements with a speed of approximately between 2.5 and 4 centimeters per second over the area of the MTP1 of the upper trapezius affected during 6 minutes.

Assessment:

To assess the effectiveness of these techniques, several tests will be performed on the subjects:

* Myotonometric measurements using a myotonometer to obtain frequency, decrement (elasticity) and stiffness of the evaluated points and MTPs.
* Algometry results will bring information of the PPT of evaluated MTPs.
* The 0-10 Numeric Pain Rating Scale results will bring information of the subjective dolor perception of the subjects.
* Inclinometer results will bring information of the ROM of cervical spine lateral inclination.
* The Neck Disability Index results will provide information on how much neck pain interferes in the daily activities of patients.

ELIGIBILITY:
Inclusion Criteria:

* Older than 18 years
* Presence of an active or latent MTrP 1 in the upper trapezius:

  * Presence of taut band in a skeletal muscle.
  * Presence of a hypersensitive point in the taut band.
  * Local twitch response caused by palpation of the taut band.
  * Reproduction of the typical referred pain pattern of MTrPs in response to compression.
  * Spontaneous presence of the typical pain pattern and/or patient's recognition of that pain as familiar (criteria only applicable to the active MTrPs).

Exclusion Criteria:

* History of neurological disorders (radiculopathy).
* Cervical surgery.
* Chronic pain in any part of the body as a result of a traumatic incident.
* Chronic rheumatic disease.
* Medical diagnosis of fibromyalgia.
* Systemic diseases.
* Actual pregnancy.
* Clinical depression.
* Body mass index ≥30.
* To receive treatment of myofascial syndrome in the muscles of the cervico-dorsal area (physical therapy, invasive techniques ...) during the month prior to the beginning of the study.
* Ingestion of medication (analgesics, muscle relaxants, psychotropic or anti-inflammatory agents) in the three days prior to the start of the study.

Exit criteria:

* Patient´s petition.
* Appearance of any lesion that might contraindicate the use of electrotherapy techniques.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2017-10-01 (Actual); Study Completion 2017-10-15 (Actual)

PRIMARY OUTCOMES:
Change in Stiffness | Pre-intervention; Post-intervention (30 minutes after intervention); Follow up (1 week after the intervention).
  The muscle stiffness reflects muscle resistance to the force that changes its shape (Nm). This outcome measure is obtained by a device named MyotonPro®. It is a non-invasive commercial device made to calculate myotonometric properties of the muscle.
Change in Decrement (elasticity) | Pre-intervention; Post-intervention (30 minutes after intervention); Follow up (1 week after the intervention).
  Logarithmic decrement of the dampening of muscle oscillations is an indicator of the elasticity. This outcome measure is obtained by a device named MyotonPro®. It is a non-invasive commercial device made to calculate myotonometric properties of the muscle.
Change in Frequency | Pre-intervention; Post-intervention (30 minutes after intervention); Follow up (1 week after the intervention).
  Frequency of muscle oscillations (Hz) is an indicator of the tone. This outcome measure is obtained by a device named MyotonPro®. It is a non-invasive commercial device made to calculate myotonometric properties of the muscle. The assessment is realized in these points:
  * MTrP 1 of the affected superior trapezius.
  * MTrP 3 of the affected superior trapezius.
  * MTrP 1 of the NO affected superior trapezius.
  * Point in the middle of the muscle belly of the affected superior trapezius. 10 mechanical stimuli of 0.4 N of force and 0.15 ms of duration will be applied. The MyotonPro® must remain perpendicular to the surface to be measured (the subject will be lying in a prone position for the MTrP 3, and sit down for the three other points). Each assessment will consist of 10 multiple measurements, spaced for 1 second. To be considerate as valid, the variation coefficient of the measure should not exceed 3%.

SECONDARY OUTCOMES:
Change in the Pressure Pain Threshold (PPT) | Pre-intervention; Post-intervention (30 minutes after intervention); Follow up (1 week after the intervention).
  The PPT is measured using a pressure algometer in these points:
  * MTrP 1 of the affected superior trapezius.
  * MTrP 3 of the affected superior trapezius.
  * MTrP 1 of the NO affected superior trapezius.
  * MTrP 2 of the lateral gastrocnemius of the affected side. The subject will be lying in a prone position for more stability and with a pillow under his feet. The algometer must remain perpendicular to the surface to be measured. It will be measured three consecutive times, with an interval of 30 seconds between each measurement.
Change in the Range Of Motion (ROM) of cervical spine lateral inclination | Pre-intervention; Post-intervention (30 minutes after intervention); Follow up (1 week after the intervention).
  It will be used a portable inclinometer to assess the ROM of the contralateral active cervical spine inclination. The subject will be in a relaxed and comfortable sitting position, leaning on the backrest, arms resting on his knees and fixing a point with his eyes. It will be measured three consecutive times, with an interval of 30 seconds between each measurement.
Change in Pain Perception | Pre-intervention; Post-intervention (30 minutes after intervention); Follow up (1 week after the intervention).
  Change in pain perception using Numeric Pain Rating Scale (NPRS). The NPRS is a scale from 0-10 ("0" = no pain; "10" = the most intense pain imaginable).
Change in Neck Disability Index (NDI) | Pre-intervention; Follow up (1 week after the intervention).
  The NDI consists of ten questions in the following domains: Pain Intensity, Personal Care, Lifting, Reading, Headaches, Concentration, Work, Driving, Sleeping, and Recreation.

CONTACTS AND LOCATIONS:
Overall Officials: Carolina Jiménez-Sánchez, MSc, Principal Investigator — Universidad San Jorge; Maria Ortiz-Lucas, PhD, Principal Investigator — Universidad San Jorge
Locations (1):
- Universidad San Jorge, Villanueva de Gállego, Spain

IPD SHARING:
Plan to Share IPD: No